CLINICAL TRIAL: NCT00904761
Title: Effects of Physical Training on Heart Rate Variability and Exercise Capacity in Diabetes With Autonomic Neuropathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 25670
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2012-12-28 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; autonomic neuropathy; exercise training; exercise capacity; heart rate variability
MeSH Terms: conditions — Diabetes Mellitus | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Experimental): arm: intervention
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — The exercise group took supervised aerobic training twice per week at hospital and thrice per week at home for eight weeks at the intensity of 60-70% VO2peak

SUMMARY:
This study aimed to investigate effects of physical training on exercise capacity and changes of heart rate variability (HRV) at rest, during exercise, and post-exercise in the patient with diabetes with autonomic neuropathy (DAN).

ELIGIBILITY:
Inclusion Criteria:

* aged under 65 years old
* receiving regular treatment
* HbA1c < 8.0
* decreased HR response in deep breathing maneuver

Exclusion Criteria:

* heart disease
* neuro-musculo-skeletal diseases
* taking any medication that may affect HRV (such as α or β-blockers)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2002-05 (Actual); Study Completion 2002-05 (Actual)

PRIMARY OUTCOMES:
heart rate variability | 8 weeks
exercise capacity | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, Doctor, Study Director — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan